CLINICAL TRIAL: NCT06681428
Title: A Multi-Center, Randomized Controlled Clinical Investigation Evaluating an Amnion/Chorion/Amnion Allograft, Amnion/Chorion Allograft, And/or an Amnion/Amnion Allograft Versus Standard of Care in the Treatment of Non-Healing Diabetic Foot Ulcers
Brief Title: Rising Tide - Amniotic Tissue(s) Treatments for Chronic Diabetic Foot Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tides Medical (Industry)
Collaborators: Professional Education and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TID-ART-01
Record Dates: First submitted 2024-11-04; First posted 2024-11-08 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Foot Ulcer (DFU); Chronic Foot Ulcers
Keywords: Amnion; Chorion; Amnion Amnion Graft; Amnion Chorion Amnion Grafts; Amnion Chorion Graft; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Pathologic Processes; Ulcer; Skin Ulcer; Chronic Ulcer; Chronic Foot Ulcer; Diabetic Angiopathies; Diabetes Type 2; Diabetes Type II; Leg Ulcer; Placental-Based Allografts; Human Placental-Based Skin Grafts; Skin Wound Covering
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Pathologic Processes; Ulcer; Skin Ulcer; Diabetic Angiopathies; Diabetes Mellitus, Type 2; Leg Ulcer | interventions — Transplantation, Homologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- "Amnion/Chorion/Amnion" common/general allograft configuration (Experimental): Topical application of placental allograft on to surface of open chronic diabetic foot ulcer using a tri-layer dehydrated amniotic membrane allograft for the treatment of DFUs. Human amniotic membrane is a thin collagenous membrane derived from the submucosa of the placenta, the organ that connects the developing fetus to the mother's uterus. A human amniotic membrane consists of multiple layers including epithelial cells, a basement membrane, and a stromal matrix which provides a natural scaffold that allows cellular attachment or infiltration and growth factor storage.
  Interventions: Other: Allograft
- Standard of Care (No Intervention): Standard of Care (SOC) for open chronic diabetic foot ulcer using a calcium alginate dressing and will have a silicone non-adherent dressing (MepitelTM or equivalent), a padded 3-layer dressing comprised of 4x4 gauze pads, soft roll, compressive wrap and Coban (Threeflex 3-layer or equivalent) applied. Offloading of the DFU (removable offloading boot or total contact casting [TCC] if the subject's foot is too large for a removable offloading boot), appropriate sharp or surgical debridement, and infection management. Graft provides a protective cover and supports the body's wound healing processes. This allograft is supplied sterile and not intended to be removed.
- "Amnion/Chorion" common/general allograft configuration (Other): Topical application of placental allograft on to surface of open chronic diabetic foot ulcer using a dehydrated human amniotic membrane allograft comprised of a tri-layer membrane (amnion/intermediate layer/chorion) which provides a natural scaffold that allows cellular attachment and infiltration. Human amniotic membrane is a thin collagenous membrane derived from the submucosa of the placenta. A human amniotic membrane consists of multiple layers including epithelial cells, a basement membrane, and a stromal matrix. Graft provides a protective cover and supports the body's wound healing processes. This allograft is supplied sterile and not intended to be removed.
  Interventions: Other: Allograft
- "Amnion/Amnion" common/general allograft configuration (Other): Topical application of placental allograft on to surface of open chronic diabetic foot ulcer using a dual layer dehydrated human amniotic membrane allograft. Human amniotic membrane is a thin collagenous membrane derived from the submucosa of the placenta, the organ that connects the developing fetus to the mother's uterus. A human amniotic membrane consists of multiple layers including epithelial cells, a basement membrane, and a stromal matrix which provides a natural scaffold that allows cellular attachment or infiltration and growth factor storage. This allograft provides a protective cover and supports the body's wound healing process. This allograft is supplied sterile and not intended to be removed.
  Interventions: Other: Allograft

INTERVENTIONS:
Other: Allograft — Placental-based Allografts
  Arms: "Amnion/Amnion" common/general allograft configuration; "Amnion/Chorion" common/general allograft configuration; "Amnion/Chorion/Amnion" common/general allograft configuration

SUMMARY:
The purpose of this clinical investigation is to evaluate the safety and efficacy of Amnion/Chorion/Amnion allograft , Amnion/Chorion allograft, and/or Amnion/Amnion allograft, plus Standard of Care (SOC) each versus SOC alone in the treatment of chronic non-healing diabetic foot ulcers (DFU) after 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects are required to meet all of the following criteria for enrollment into the study.

1. At least 18 years old, inclusive.
2. Presence of a DFU, Wagner Grade 1, extending through the dermis provided it is below the medial aspect of the malleolus.
3. The index ulcer (ulcer to be evaluated in the study) will be the largest ulcer if two or more DFUs are present with the same Wagner grade and will be the only one evaluated in the study. If other ulcerations are present on the same foot, they must be more than 2 cm distant from the index ulcer.
4. Index ulcer has been present for greater than 4 weeks prior to SV1 and less than 1 year, as of the date the subject consents for study.
5. Index ulcer is a minimum of 1.0 cm2 and a maximum of 25 cm2 at SV1 and TV1.
6. Within 3 months of SV1, adequate circulation to the affected foot as documented by a dorsal transcutaneous oxygen measurement (TCOM) or a skin perfusion pressure (SPP) measurement of ≥ 30 mmHg, or an Ankle Branchial Index (ABI) between 0.7 and 1.3 using the affected study extremity. As an alternative, arterial Doppler ultrasound can be performed evaluating for biphasic dorsalis pedis and posterior tibial vessels at the level of the ankle or a TBI (Toe Brachial Index) of > 0.6 is acceptable.
7. The target ulcer has been offloaded for at least 14 days, prior to TV1.
8. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers or abstinence) during the course of the study and undergo pregnancy tests.
9. Subject understands and is willing to participate in the clinical study and can comply with weekly visits.
10. Subjects must have read and signed the IRB approved ICF before screening procedures are performed.

Exclusion Criteria:

Potential subjects meeting any of the following criteria will be excluded from enrollment and subsequent treatment.

1. Index ulcer(s) deemed by the investigator to be caused by a medical condition other than diabetes
2. Index ulcer, in the opinion of the investigator, is suspicious for cancer and should undergo an ulcer biopsy to rule out a carcinoma of the ulcer
3. Index ulcer is infected
4. Subjects with a history of more than two weeks of treatment with immune-suppressants (including systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within 1-month prior to first SV1, or who receive such medications during the screening period or who are anticipated to require such medications during the course of the study
5. Subjects on any investigational drug(s), Investigational products, or therapeutic device(s) within 30 days preceding SV1
6. History of radiation at the ulcer site (regardless of time since last radiation treatment)
7. Index ulcer has been previously treated or will need to be treated with any prohibited therapies
8. Subjects with a previous diagnosis of HIV or Hepatitis C
9. Presence of any condition(s) which seriously compromises the subject's ability to complete this study or has a known history of poor adherence with medical treatment
10. Osteomyelitis or bone infection of the affected foot as verified by x-ray within 30 days prior to the first screening visit. (In the event of an ambiguous diagnosis, the Principal Investigator will make the final decision)
11. Subject is pregnant or breast-feeding
12. Presence of diabetes with poor metabolic control as documented with an HbA1c >12.0 within last 90 days
13. Subjects with end stage renal disease as evidenced by a serum creatinine ≥3.0 mg/dL within 6 months of enrollment
14. Presence of acute Charcot Neuroarthropathy to the affected limb
15. Index ulcer that has reduced in area by 30% or more after 14 days of SOC from SV1 to the TV1/Randomization visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2026-11-18 (Estimated); Study Completion 2026-11-18 (Estimated)

PRIMARY OUTCOMES:
Percentage of DFUs healed at 12 weeks | 12 Weeks
  Percentage of index ulcers (the ulcers being treated in the study) healed at 12 weeks

SECONDARY OUTCOMES:
Total time to DFU wound closure | 12 Weeks
  Length of time to complete wound closure of the indexed DFU
Percentage of Wound Area Reduction over time of study | 12 Weeks
  Percentage area reduction by surface area for each indexed wound during the clinical investigation
Change in perceived patient wound pain levels over time. | 12 weeks
  Change in patient pain levels during the clinical investigation at the wound site using the pain assessment by questionnaire. The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

OTHER OUTCOMES:
Cost of Treatment to Closure Diabetic Foot Ulcer Wound in Study | 12 Weeks
  Following costs to treat and closure diabetic foot ulcers in investigational study arms

CONTACTS AND LOCATIONS:
Overall Officials: David G Armstrong, DPM, MD, PhD, Study Chair — Keck School of Medicine of USC; Frank Burrows, MBA, EMT, BCMAS, CWCA, Study Director — Tides Medical
Locations (9):
- United States (9):
  - Limb Preservation Platform Inc, Fresno, California
  - Angel City Research, Los Angeles, California
  - Clemente Clinical Research, Los Angeles, California
  - ILD Research Center, Vista, California
  - Clever Medical Research, Miami, Florida
  - Foot and Ankle Specialists of the Mid-Atlantic, Raleigh, North Carolina
  - Lower Extremity Institute of Research and Therapy, Boardman, Ohio
  - Brock Liden DPM, Circleville, Ohio
  - Foot and Ankle Specialists of the Mid-Atlantic, Salem, Virginia

IPD SHARING:
Plan to Share IPD: Undecided